CLINICAL TRIAL: NCT01618877
Title: A Monocenter, Open-label, Two-way Randomized Cross-over Study to Evaluate the Bioequivalence of Levetiracetam Administered as a 45 Minutes Intravenous Infusion and Same Dosage Levetiracetam Oral Tablet (Part A); and a Randomized, Double-blind, Placebo-controlled, Parallel Study on the Safety, Tolerability and Pharmacokinetics of Levetiracetam 45 Minutes Intravenous Infusion During 4 Days of b.i.d. Dosing (Part B), in Chinese Healthy Volunteers
Brief Title: A Randomized, Double-blind, Pharmacokinetics Study to Assess Safety, Tolerability of Levetiracetam 45 Minutes Intravenous Infusion During 4 Days of Bid Dosing in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01362B
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Human Volunteers
Keywords: Keppra Levetiracetam intravenous; Multiple dose; Safety; Pharmacokinetics; Chinese healthy volunteers
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam iv infusion (Experimental): Levetiracetam intravenous (iv) infusion.
  Interventions: Drug: Levetiracetam
- Placebo infusion (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levetiracetam — Levetiracetam 1.500 mg (500 mg/ 5 mL vials) administered as a 45 minutes intravenous infusion diluted in 100 mL 0.9 % saline solution every 12 hours from the morning of Day 3 (it is the first day in Part B) to the morning of Day 7 (it is the 5th day in Part B).
  Other Names: Keppra
  Arms: Levetiracetam iv infusion
Other: Placebo — 15 mL 0.9 % saline solution added to 100 mL 0.9 % saline solution, administered as a 45 minutes intravenous infusion every 12 hours from the morning of Day 3 ( it is the 1st day in Part B) to the morning of Day 7 (it is the 5th day in Part B).
  Arms: Placebo infusion

SUMMARY:
The part B of N01362 is to assess the pharmacokinetic profile of Levetiracetam 1500 mg intravenous (iv) infusion during repeated dosing in Chinese healthy volunteers.

DETAILED DESCRIPTION:
The study includes 2 parts, part A is to evaluate the bioequivalence of Levetiracetam (LEV) 1500 mg intravenous (iv) infusion when compared to oral tablet, part B is to assess the pharmacokinetic profile of LEV infusion during repeated dosing in Chinese healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Chinese, age 18-40, weight ≥ 50 kg
* Healthy volunteers with normal vital signs, good physical and mental health status and normal electrocardiogram and laboratory test

Exclusion Criteria:

* History or presence of each systems disorders capable of altering the absorption, metabolism or elimination of drugs, or of constituting a risk factor when taking the study medication
* History or presence of drug addiction or excessive use of alcohol
* Symptomatic or asymptomatic Orthostatic Hypotension at screening
* Current smokers and former smokers
* Heavy caffeine drinker
* History of frequent and severe headache
* Any drug treatment
* Subjects who are known to have Serum Hepatitis or who are carriers of the Hepatitis B surface antigen, or Hepatitis C antibody or who are HIV positive
* Subjects on a controlled sodium diet
* Subject has made a blood donation or had a comparable blood loss

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve over a dosing interval (AUCτ) | Pharmacokinetic samples were taken 36 hours after iv administration on Day 7
  The AUCτ is the area under the plasma concentration, after the last intravenous (iv) dose, versus time curve observed during the dosing interval τ.
Maximum measured plasma concentration (Cmax) | Pharmacokinetic samples were taken 36 hours after iv administration on Day 7
  The value of the maximum plasma concentration is directly obtained from the observed plasma concentration versus time curves.

SECONDARY OUTCOMES:
Plasma concentration at the end of the 45-minutes intravenous (iv) infusion (C45'(iv)) | Pharmacokinetic samples were taken 36 hours after iv administration on Day 7
  The value of the plasma concentration at the end of the 45-min iv infusion is directly obtained from the experimental data of plasma concentration versus time curves.
Minimum plasma concentration over dosing interval after intravenous (iv) infusion (Cmin) | Pharmacokinetic samples were taken 36 hours after iv administration on Day 7
Terminal half-life (t1/2) | Pharmacokinetic samples were taken 36 hours after iv administration on Day 7
  The terminal half-life associated with the terminal rate constant λ_z is calculated as: ln2/λ_z. λ_z is the first order rate constant of elimination.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- 1, Shanghai, China

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm